CLINICAL TRIAL: NCT03053687
Title: Effect of Nutritional Formula Supplementation on Growth Rate of Growth Hormone (GH) Treated Children With Growth Hormone Deficiency (GHD) After the Second Year of Therapy- a Randomized Double Blind, Placebo Controlled Trial
Brief Title: Effect of Nutritional Formula Supplementation on Growth Rate of Growth Hormone (GH) Treated Children With Growth Hormone Deficiency (GHD) After the Second Year of Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rmc082116ctil
Record Dates: First submitted 2017-02-07; First posted 2017-02-15 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: IGHD - Isolated Growth Hormone Deficiency; Growth Retardation
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional Standardized Supplementation Formula (Experimental): Powder added to water, containing about 25% of recommended Daily Recommended Intake (DRI) for calories, high protein (25% of calories) and multivitamin and mineral (25%-100% of DRI for recommended daily allowance (RDA) or adequate intake
  Interventions: Dietary Supplement: Nutritional supplementation standardized formula
- Placebo (Placebo Comparator): Low caloric formula (Powder added to water) without added vitamins and mineral
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nutritional supplementation standardized formula — Powder added to water, containing about 25% of recommended Daily Recommended Intake (DRI) for calories, high protein (25% of calories) and multivitamin and mineral (25%-100% of DRI for recommended daily allowance (RDA) or adequate intake
  Arms: Nutritional Standardized Supplementation Formula
Dietary Supplement: Placebo — Low caloric formula (Powder added to water) without added vitamins and mineral
  Arms: Placebo

SUMMARY:
The Proposed study is a double blind, randomized, placebo controlled study The aim of the study is to evaluate the effect of combined Growth Hormone (GH) treatment & nutritional formula supplementation versus GH & placebo on growth parameters in 64 children with Isolated Growth Hormone Deficiency (IGHD) after the 2nd year of GH treatment.

In this trial GH is a background treatment (non-investigational medicinal product. Participants may be treated with any of the commercial GH products approved in Israel for the indication of IGHD.

Participants will be randomly assigned either to the intervention group or the placebo control group. Randomization for the two study groups will be made in a ratio of 1:1. Both participants and study team will be blinded to the type of treatment that each patient will receive during the study. The randomization will be done according to gender and tanner stage.

Participants in the intervention groups will be treated with the study formulas and participants in the control group will be treated with a placebo low caloric formulas (Powder added to water) The study will continue for 6 months of intervention versus active placebo, with additional 6 months (an extension period), in which participants at both groups, the intervention and the placebo, will be offered to continue their participation in the study with the active study supplement.

ELIGIBILITY:
Inclusion Criteria:

* GH treatment for at least 24 months due to IGHD. Confirmed diagnosis of GHD as determined by at least one GH stimulation test, defined as a peak GH level of ≤ 10 ng/ml
* Boys: testicular volume < 8ml; Girls: breast ≤ Tanner 3
* weight SDS < 0
* BMI SDS < 50 precentile for age and gender
* Signing inform consent forms

Exclusion Criteria:

* Other indication for GH treatment.
* Bone age: boys>13.5, girls>11.5.
* Any known morbidity: chronic disease dysmorphic syndromes, bone diseases, organic brain diseases, neurological disease, past or current malignancy, chronic cardiac, renal or pulmonary problems, metabolic disorders.
* Any known gastrointestinal problem including absorption problems.
* Any chronic treatment with medication that might affect appetite, weight or growth (for example steroids) except from Ritalin use
* Any eating disorders and/or psychiatric disorder

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Weight Standard Deviation Score (SDS) | at 6 months

SECONDARY OUTCOMES:
Height-SDS | at 12 months
Weight SDS | at 12 months
BMI SDS | at 12 months

OTHER OUTCOMES:
Body composition | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, MD, Principal Investigator — Schneider Children's Medical Center
Locations (1):
- Schnider children's medical center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No